CLINICAL TRIAL: NCT04395261
Title: The Differential Diagnosis of Different Middle Ear Fluids in Otitis Media With Effusion by Wideband Tympanometry
Brief Title: Wideband Tympanometry in Otitis Media With Effusion
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Prof.Dr., Pamukkale University
Other Study IDs: 3
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Otitis Media With Effusion
MeSH Terms: conditions — Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 0: Patients were divided into groups according to observation in surgery Empty ear in operation
  Interventions: Diagnostic Test: Wideband Tympanometry
- Group 1: Patients were divided into groups according to observation in surgery Serous fluid in operation
  Interventions: Diagnostic Test: Wideband Tympanometry
- Group 2: Patients were divided into groups according to observation in surgery Mucoid fluid in operation
  Interventions: Diagnostic Test: Wideband Tympanometry
- Group 3: Patients were divided into groups according to observation in surgery Adhesive tympanic membrane in operation
  Interventions: Diagnostic Test: Wideband Tympanometry
- Group 4: Control group. Subjects with no otitis media with effusion
  Interventions: Diagnostic Test: Wideband Tympanometry

INTERVENTIONS:
Diagnostic Test: Wideband Tympanometry

SUMMARY:
The investigators asked the question if they can better estimate the middle ear status in OME that help them to decide between early intervention or longer follow up.

DETAILED DESCRIPTION:
Purpose: Otitis media with effusion is an important problem in childhood. After proper diagnosis, generally 3 months of follow up has been recommended before surgical tympanostomy tube insertion. If the physician can estimate the status of the middle ear or fluid type better with a non-invasive method, we can suggest an early operation to these patients or decide to follow up more with no intervention. The purpose of the study is to compare the surgically confirmed middle ear effusions with wideband absorbance values and to differentiate them noninvasively before the operation.

Methods: A total of 123 children that were followed 3 months and treated surgically with the diagnosis of OME were included. Eighty-two sex, age-matched children were tested as control with wideband tympanometry. Ears were divided into four groups according to findings in the operation: serous, mucoid, adhesive, empty. Resonance frequency, 226 Hz, 1000 Hz compliance, Wideband Peak pressure, Absorbance measurements used for comparison.

ELIGIBILITY:
Inclusion Criteria:

* All patients were diagnosed by ear examination, pneumatic otoscopy, and type B tympanogram with 226 Hz tympanometry. They were followed for 3 months with proper medication. After 3 months if there was no change with ear examination and 226 Hz tympanometry, surgical ventilation tube insertion was offered.

Exclusion Criteria:

* The patients with chronic ear diseases, ototoxic drug use, neurologic disease were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: children with otitis media with effusion
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Resonance frequency | The same 1 day with the operation
  Wideband resonance frequency was measured
Absorbance | The same 1 day with the operation
  Wideband absorbance of frequencies between 250-8000 Hz were measured

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Chief of Department

IPD SHARING:
Plan to Share IPD: No
Data will be available in the university depository